CLINICAL TRIAL: NCT01202578
Title: A Clinical Study of the Acclarent Tympanostomy Tube Delivery System for the Treatment of Patients Requiring Tympanostomy Tube Insertion for Otitis Media
Brief Title: Evaluation of the Tympanostomy Tube Delivery System
Acronym: inVENT-OR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005013
Record Dates: First submitted 2010-09-13; First posted 2010-09-16 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media With Effusion; Acute Otitis Media
MeSH Terms: conditions — Otitis Media with Effusion; Otitis Media | interventions — Middle Ear Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tympanostomy tube (Experimental): performance and safety of tympanostomy tube delivery system
  Interventions: Device: tympanostomy tube

INTERVENTIONS:
Device: tympanostomy tube — tympanostomy tube delivery system

SUMMARY:
The purpose of this study is to evaluate the performance and safety of the Tympanostomy Tube Delivery System (TTDS) for chronic otitis media or recurrent acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either chronic otitis media with effusion or acute otitis media and scheduled to undergo tympanostomy tube insertion

Exclusion Criteria:

* Reaction to anesthesia
* Markedly atrophic, bimeric, severely retracted, atelectatic or perforated tympanic membrane
* Otitis externa
* Active acute otitis media
* Otitis media pathology requiring T-tubes
* Stenosed ear canal
* Anatomy that precludes visualization and access to tympanic membrane
* Anatomy that necessitates tympanostomy tube placement in posterior half of membrane

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Faw, MD, Principal Investigator — Evergreen Sinus Center; Andrew Gould, MD, Principal Investigator — Advanced ENT and Allergy; Charles Syms, MD, Principal Investigator — Ear Medical Group; Jacob Zeiders, MD, Principal Investigator — South Coast ENT
Locations (4):
- United States (4):
  - South Coast ENT, Port Saint Lucie, Florida
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Ear Medical Group, San Antonio, Texas
  - Evergreen Sinus Center, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects presenting to the clinical study site for whom tympanostomy tube insertion was recommended were offered the opportunity to participate in the study by study investigators.
Period: Overall Study
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.68 (2.49)
Age, Customized [Number; unit: participants]
  <=5 years | 47
  >5 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Safety of Tympanostomy Tube (TT) Delivery System
Description: Occurrence of pre-defined Safety Events of acoustic trauma, deployment of the TT into the middle ear, damage to middle ear structures, unintended tympanic membrane perforation requiring treatment, abrasion to the external acoustic meatus requiring significant treatment, and major bleeding requiring significant treatment.
Time Frame: 7 days
Population: Subjects in whom TTDS was attempted.
Measure: Number (95% Confidence Interval); unit: percentage of ears
Units Other Than Participants: ears
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Number analyzed (Participants) | 53
Number analyzed (ears) | 101
percentage of ears | 0.0 [0.0 to 3.6]

2. Primary Outcome: Device Success
Description: Device Success is defined as the successful delivery of the tympanostomy tube across the tympanic membrane using the tympanostomy tube delivery system (TTDS).Device Success is evaluated on a per device basis.
Time Frame: 0 days
Population: Device Success is evaluated on a per device basis.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: devices
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Number analyzed (Participants) | 53
Number analyzed (devices) | 101
percentage of devices | 94.1 [87.5 to 97.8]

3. Secondary Outcome: Proportion of Subjects With Procedure Success
Description: Procedure Success was defined as the successful placement of any tympanostomy tube in all enrolled ears in a given subject. Non-Acclarent tubes successfully placed manually following non-success of the TTDS were counted toward Procedure Success. Procedure Success was determined on a per subject basis: the rate was calculated by the number of subjects achieving Procedure Success out of the total number of enrolled subjects.
Time Frame: 0 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Number analyzed (Participants) | 53
percentage of participants | 100 [93.3 to 100.0]

4. Secondary Outcome: Tube Retention
Description: Presence of the tympanostomy tube across the tympanic membrane at the follow-up visit.
Time Frame: 7 days
Population: Tube retention was assessed for all TT successfully placed by the TTDS
Measure: Number (95% Confidence Interval); unit: percentage of tubes retained
Units Other Than Participants: tympanostomy tubes placed by TTDS
Arm/Group | Tympanostomy Tube Placement Using the Tube Delivery System
Number analyzed (Participants) | 53
Number analyzed (tympanostomy tubes placed by TTDS) | 95
percentage of tubes retained | 99.0 [94.3 to 100.0]

ADVERSE EVENTS:
Time Frame: 7 days
Description: Adverse events occured only in study cohort (non lead-in) participants.
Groups:
- Safety Events: Safety in terms of number affected subjects in total number of subjects.
Arm/Group | Safety Events
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 4/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Events (N=53)
Tube Lumen Occlusion (Ear and labyrinth disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days